CLINICAL TRIAL: NCT00035373
Title: Eligibility Screening of Patients With Central Nervous System Tumors for the National Cancer Institute (NCI) Clinical Research Protocols
Brief Title: Eligibility Screening of Patients With Central Nervous System Tumors for the National Cancer Institute s (NCI) Clinical Research Protocols
Status: Terminated | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020186; 02-C-0186; NCT00040924 (obsolete NCT alias)
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2015-04-29

CONDITIONS: Glioblatoma; Gliosarcoma; Anaplastic Astrocytoma; Oligodendroglioma; Anaplastic Oligoastrocytoma
Keywords: Tumor; Brain; Chemotherapy; Anti-Angiogenesis; Radiation Therapy; CNS Tumor
MeSH Terms: conditions — Gliosarcoma; Astrocytoma; Oligodendroglioma; Neoplasms; Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The objective of this study is to evaluate patients with tumors of the central nervous system (CNS) for eligibility in the National Cancer Institute s research studies. These patients will undergo a series of procedures, usually including a complete medical history and physical examination; laboratory testing of blood, CSF, urine, bone marrow, or other samples; an evaluation of tumor location and size by x-rays, CT (computed tomography) or MRI (magnetic resonance imaging) scans, or nuclear medicine scans; lumbar puncture; electrocardiogram and echocardiogram; and procedures to evaluate the function of specific organs. A bone marrow biopsy is occasionally performed. Research samples may also be collected and stored to avoid having to do a painful test more than once. Tissue specimens collected during this process may be stored and used in future studies.

Patients of both genders, any age, and all racial and ethnic groups with tumors of the CNS or a history of a CNS tumor are eligible. Up to 100 people are expected to participate.

The physician will discuss the results of these procedures with the patient and his or her family. On the basis of the eligibility screening and the patient s wishes, the patient may then be enrolled in a primary research protocol.

DETAILED DESCRIPTION:
BACKGROUND:

-Adult patients (greater than or equal to 18 yrs of age) with tumors of the central nervous system who are being evaluated by the Neuro-Oncology Branch (NOB) for National Cancer Institute (NCI) primary research protocols will be entered onto this screening protocol for eligibility screening.

OBJECTIVE:

- Evaluate patients with tumors of the Central Nervous System (CNS) for eligibility in National Cancer Institute (NCI) research protocols.

ELIGIBILITY:

- Patients with tumors of the CNS or a history of a CNS tumor who are being evaluated for protocols within the National Cancer Institute.

DESIGN:

* The screening tests and procedures that are required by the primary research protocols will be conducted in order to establish eligibility for these protocols.
* These procedures may include, but are not limited to, laboratory tests on blood, CSF, urine, or other specimens, and radiographic and nuclear medicine studies, which may require the administration of contrast or a radioisotopic tracer.
* This protocol will also allow for evaluation of existing tumor specimens to determine if targets are present, when applicable.
* In some cases, specific research samples required for the primary research protocol may be collected during the screening process in order to prevent us from having to subject the patient to a painful procedure on multiple occasions (e.g., bone marrow aspirations).
* Research specimens will be discarded, if the patient is not eligible for or elects not to enroll on the primary research protocol. A total of 3000 patients will be enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adult patients (greater than or equal to 18 yrs of age) with tumors of the CNS or a history of a CNS tumor who are being evaluated for protocols within the National Cancer Institute.

All patients or their previously designated LAR (Legally Authorized Representative) (if the patient is deemed by the treating physician to be impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable) must sign an informed consent indicating that they are aware of the investigational nature of this study and the risks of the procedures that will be performed to assess eligibility for primary research protocols.

EXCLUSION CRITERIA:

None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 767 (Actual)
Dates: Start 2002-04-19; Study Completion 2015-04-29

PRIMARY OUTCOMES:
Evaluate patients with tumors of the Central Nervous System (CNS) for eligibility in National Cancer Institute (NCI) research protocols. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Warren, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States